CLINICAL TRIAL: NCT05307393
Title: Maternal Positioning to Correct Fetal Occiput Posterior in the First Stage of Labor
Brief Title: Maternal Positioning to Correct Fetal Occiput Posterior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-0519
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Obstetric Complication
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (No Intervention)
- B (Experimental): Group B will be placed in a dorsal recumbent, modified sims position on the side of fetal movement.
  Interventions: Behavioral: Positioning
- C (Experimental): Group C, will be placed in the same position but opposite that of which fetal kicks are felt.
  Interventions: Behavioral: Positioning

INTERVENTIONS:
Behavioral: Positioning — Upon admission to labor and delivery, following an initial ultrasound to confirm fetal OP position, women in this study will be randomly assigned to one of three groups; one control (Group A), and two experimental (Groups B and C) groups. Those assigned to Group A will be allowed to remain in any position they chose during their labor and delivery course. Group B will be placed in a dorsal recumbent, modified sims position on the side of fetal movement. Group C, will be placed in the same position but opposite that of which fetal kicks are felt.
  Arms: B; C

SUMMARY:
In evaluating a patient's ability to have a normal vaginal delivery, a practitioner must consider three factors. Commonly referred to as the three P's, these include Power (contractions), Passage (pelvis and soft tissue) and passenger (baby). Power can be controlled through induction and augmentation agents. Passage is determined by the women's body habitus. Passenger includes the baby's estimated fetal weight (EFW) and position. Throughout the history of obstetrics, the baby's position has been a factor that has acted as a strong predictor of a woman's ability to deliver vaginally. Several researchers have looked into the percentage of babies born in the Occiput Anterior (fetus facing down) vs. Occiput Posterior (fetus facing up aka "sunny side up") position. Studies have shown that the majority of babies are born in OA position and that the finding of an OA positioned baby is associated with a greater likelihood of a successful vaginal delivery. OP position is associated with higher risk of 3rd and 4th degree perineal lacerations, operative delivery (vacuum/forceps) and cesarean section. Therefore OP position poses a higher risk of morbidity to the patient and fetus. Multiple studies exist in the obstetrics and midwifery literature regarding maternal positioning to correct fetal malposition. Many of these studies have shown no significance and those that do have generated conflicting results and are consistently lacking in power. The aim of this prospective study is to determine if maternal positioning to either the side of fetal movement (contralateral/opposite to the fetal spine) or opposite of the side of fetal movement (ipsilateral to the fetal spine) during the first stage of labor is associated with correction of fetal OP to OA position. Upon admission to labor and delivery, following an initial ultrasound to confirm fetal OP position, women in this study will be randomly assigned to one of three groups; one control (Group A), and two experimental (Groups B and C) groups. Those assigned to Group A will be allowed to remain in any position they chose during their labor and delivery course. Group B will be placed in a dorsal recumbent, modified sims position on the side of fetal movement. Group C, will be placed in the same position but opposite that of which fetal kicks are felt. Subjects in the experimental group will be asked to remain in these positions throughout the majority of their labor and delivery course, up until the second stage of labor (10 cm dilated). They will be allowed to change positions for up to 10 min per hour for maternal comfort and any fetal resuscitation efforts. Anything longer than this will be considered a deviation from the protocol and will be documented as such, but all necessary intervention for fetal well-being will be allowed including changes in maternal position for longer than 10 minutes. Once a cervical dilation of 10cm is achieved all study interventions will be discontinued. Peanut balls and manual rotational maneuvers will not be allowed as they are considered confounding factors which may individually affect fetal position. Data will be collected from the hospital record. This data will include: maternal age, BMI, race, maternal medical complications, delivery type, laceration, fetal position at delivery, dilation on admission and weight of the baby.

ELIGIBILITY:
Inclusion Criteria:

* Women who are >/=18yo
* able to consent
* >/=37 weeks gestation (full term) with a viable singleton intrauterine pregnancy noted to be cephalic presentation in the OP position at the time of admission as noted on bedside ultrasound
* All patients must be <10cm, with a score of 3 or less out of 10 on a numeric pain rating scale
* admitted to LIJ or NSUH for either spontaneous labor or labor induction.

Exclusion Criteria:

* All women younger than 18yo
* unable to consent
* admitted in the second stage of labor (>10cm) or beyond, with nonviable pregnancies (i.e. IUFD), score of 4 or more on a numeric pain rating scale, or desiring cesarean section will be excluded.
* all women with pregnancies noted to have IUGR, fetal anomalies, malpresentation (i.e. breech), multiple gestations or fetuses not in the OP position at time of admission will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 465 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Fetal Position at time of delivery | From time of admission to delivery
  Rate of OA position in each arm at time of delivery

SECONDARY OUTCOMES:
Mode of delivery | From time of admission to delivery
  Vaginal delivery rates in each arm
Laceration Type | From time of admission to delivery
  Incidence of 3rd and 4th degree lacerations in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Schulz, MD, Principal Investigator — Northwell Health; Sarah Pachtman, MD, Principal Investigator — Northwell Health
Locations (1):
- Long Island Jewish medical center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No